CLINICAL TRIAL: NCT07197502
Title: CLINICAL TRIAL: Treatment of Borderline Personality Disorder by Targeting Ventrolateral Prefrontal-amygdala Circuit With Network-based Neuronavigated Transcranial Magnetic Stimulation
Brief Title: Treatment of Borderline Personality Disorder With rTMS
Acronym: ClinicalBPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Andrew F. Leuchter, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 23-001340
Record Dates: First submitted 2025-09-18; First posted 2025-09-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Borderline Personality Disorder; Borderline Personality; BPD - Borderline Personality Disorder
Keywords: BPD; rTMS; TMS; Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active (Experimental): Subjects in this group will receive active TMS treatment at vlPFC delivered by a magnet called A/P (active/placebo) coil. The A/P coil supports double-blinding of treatment. The coil has two sides, one of which is shielded so that no energy is imparted to the brain when the shielded side is applied to the subject's head. Small skin electrodes are applied to the scalp under the coil that impart a small microcurrent to the scalp simulating the sensation of active treatment. The operator receives a code from the device instructing them which side of the coil to use for each subject, ensuring complete treatment blinding.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham- followed by Active treatment (Experimental): Patients will be randomized to receive active or sham at vlPFC. Subjects assigned to the sham-controlled condition will be oﬀered the opportunity to cross-over to open - label TMS treatment at the conclusion of the double-blind phase. This phase will serve as an incentive to recruitment because it ensures that all subjects (even those initially receiving sham stimulation) will eventually be eligible to receive active treatment. Rating scale scores will be obtained in the open-label extension just as scheduled in the controlled phase to gather additional information on eﬃcacy of the active intervention.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transcranial magnetic stimulation (TMS) is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain to improve symptoms of depression. Using pulsed magnetic fields, transcranial magnetic stimulation therapy stimulates the part of the brain thought to be involved with mood regulation. These magnetic fields do not directly affect the whole brain; they only reach about 2-3 centimeters into the brain directly beneath the treatment coil.As these magnetic fields move into the brain, they produce very small electrical currents. These electrical currents activate cells within the brain, causing them to rewire, a process called neuroplasticity.

SUMMARY:
This project studies the effectiveness of brain stimulation on borderline personality disorder (BPD) symptoms. This study is blinded, randomized and will enroll up to 30 participants.

Participant will be consented for the study remotely via a secure internet platform called Zoom.

Participants will undergo up to 2 MRI scans, 2 brain wave recording sessions and up to 30 brain stimulation treatments, and complete symptom assessments and cognitive behavioral tasks on a computer. Participation requires minimum of 17 in person visits over the course of 2.5 months.

Participants are randomly assigned active or sham brain stimulation. Participants who received sham brain stimulation have the option to receive additional 15 active brain stimulation session.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a serious and pervasive psychiatric condition with a prevalence of 1-5% among the general population. Two core symptoms of BPD are dysfunctional emotion regulation and marked impulsivity resulting in severe psychological suffering in terms of depression and anxiety as well as maladaptive impulsive acts, particularly self-harming behaviors including suicide. Recent advances in affective neuroscience of BPD combined with progress in brain imaging and neuromodulation technologies have opened new avenues for the development of innovative, brain-based, and more effective treatments for BPD.

This project aims to test the efficacy of a novel circuit-based treatment for BPD. The investigators will utilize multimodal neuroimaging Magnetic Resonance Imaging (MRI), and electroencephalogram (EEG) and BPD-, depression- and anxiety-related clinical scales to objectively measure the impact of Transcranial Magnetic Stimulation (TMS) treatment on overall BPD as well as depressive and anxiety symptom severity. Furthermore, a battery of cognitive tasks will be used to specifically measure the effect of TMS on the neurobehavioral indicators of impulsivity and emotion regulation.

ELIGIBILITY:
* Age of 18-65
* DSM-5 Diagnosis of BPD based upon a psychiatric evaluation and ZAN-BPD
* Fluent English speaker
* Signed informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Borderline Symptom List 23 (BSL-23) | Baseline (Day 1) and Post treatment (Day 17)
  Borderline Symptom List 23 (BSL-23)
Clinical Global Impression for Borderline Personality Disorder (CGI-BPD) | Baseline (Day 1) and Post treatment (Day 17)
  Clinical Global Impression for Borderline Personality Disorder (CGI-BPD)
Diﬃculties in Emotion Regulation Scale (DERS) | Baseline (Day 1) and Post treatment (Day 17)
  Diﬃculties in Emotion Regulation Scale (DERS)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Semel Institute for Neuroscience and Human Behavior at UCLA, Los Angeles, California
  - Semel Institute/ UCLA TMS, Los Angeles, California